CLINICAL TRIAL: NCT04122157
Title: Prospective Single-center Long-term Observation of the SL-PLUS® MIA Stem
Acronym: SL-PLUS MIA
Status: Completed | Type: Observational
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Other Study IDs: D10055-2
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2021-02

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: Uncoated SL PLUS® MIA stem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Summary from initial protocol

Goal: Validation of the uncoated SL-PLUS® MIA stem within an observation study

Study design: prospective, single-center, observational, non-comparative study

Study population: 135 consecutive cases (uncoated SL-PLUS® MIA implants)

Intervention (if applicable): Implantation of a total hip endoprosthesis

Main goals/endpoints: Radiological: radiolucent lines, osteolysis, hypo- and hypertrophy of the cortex, loosening of the implant or migration; clinical: Harris Hip Score, implant-related complications, revisions; patient questionnaire (WOMAC)

Type and extent of the risks associated with the study participation as well as benefits for the patient: All patients will benefit from the hip prostheses without exception. There are no increased risks for the patients participating in the study compared to patients who do not participate. Normal, necessary follow-up exams will be performed over the course of 10 years. These follow-up exams will then be quantitatively evaluated within the scope of the study in accordance with a standardized protocol. Accordingly, the benefit for the patients from the participation in the study is currently not yet foreseeable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary hip osteoarthritis
* Patients scheduled for a first implantation
* Age at the time of surgery 40-80 years

Exclusion Criteria:

* Destruction of the acetabulum
* Deformation of the hip joint
* Deformation of the proximal femur
* Revision of failed hip endoprostheses
* Acute or recent infection of the joint or its surrounding region
* Acute or chronic systemic infections
* Marked atrophy or deformation of the upper femur
* Muscle atrophy or a neuromuscular disease
* Pathological fractures
* Per- to subtrochanteric fractures
* Conditions that would prevent secure anchoring of the hip prosthesis
* Obese patients with a BMI >35
* Patients not expected to have a successful rehabilitation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 135 consecutive cases (uncoated SL-PLUS® MIA implants)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2007-07-22 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Survival, Kaplan Meier | up to 10 years after implantation
  Survival rate: Rate of hip implants in situ after 10 years of follow-up.
Intra- und perioperative implant-related "Adverse Events" (AE) and complications until discharge | up to patient's discharge from the hospital/clinic (from surgery up to 7 days after surgery)
  Rate of hip implant experiencing intra- und perioperative implant-related "Adverse Events" (AE) and complications until discharge.
  Rate of hip implants with Adverse Events, Adverse Device Effects, Serious Adverse Events, Serious Adverse Device Effects
Postoperative AE up to 10 years after the surgery | up to 10 years after implantation
  Rate of hip implants experiencing Postoperative AE up to 10 years after the surgery Adverse Events, Adverse Device Effects, Serious Adverse Events, Serious Adverse Device Effects

SECONDARY OUTCOMES:
Radiographic changes defined as radiolucent lines, osteolysis, hypo- and hypertrophy of the cortex, loosening of the implant or migration. | up to 10 years after implantation
  Rate of hip implants with radiographic changes defined as radiolucent lines, osteolysis, hypo- and hypertrophy of the cortex, loosening of the implant or migration.
Harris Hip Score | up to 10 years after implantation
  The Harris Hip Score (HHS) is a clinician-based outcome measure frequently used for the evaluation of patients following a total hip arthroplasty.The score considers information on pain, function and range of motion. The scale ranges from 0 - 100 whereas, a higher score indicates a favorable outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Vinzenz v. Auersperg, Prim. Dr., Principal Investigator — Orthopädie LKH Steyr